CLINICAL TRIAL: NCT04686487
Title: Stereotactic Ablative Radiotherapy in Patients With Hypertrophic Obstructive Cardiomyopathy: First in Man Pilot Study
Brief Title: SterEotactic AbLative Radiotherapy in PatiEnts With HypertrophiC ObstrucTive Cardiomyopathy
Acronym: SELECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Shenghua Zhou, Professor, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOCM2018044
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Hypertrophic Obstructive Cardiomyopathy; Stereotactic Ablative Radiotherapy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Ablative Radiotherapy (Other): Stereotactic body radiation therapy delivered to the thick heart muscle at the point of obstruction
  Interventions: Procedure: stereotactic ablative radiotherapy

INTERVENTIONS:
Procedure: stereotactic ablative radiotherapy — stereotactic ablative radiotherapy by targeting high energy heavy ion beams at a specific area of the body

SUMMARY:
Hypertrophic obstructive cardiomyopathy (HOCM) is an inherited myocardial disease which leads to the muscle in the wall of the heart growing and thickening to the point that it blocks blood flow exiting the heart with increasing risk of sudden cardiac death, heart failure, and atrial fibrillation. Surgical septal myectomy and alcohol septal ablation are two invasive therapies for drug-refractory symptomatic patients with HOCM. Unfortunately, some patients may be unsuitable for both the two procedures. Recently, stereotactic ablative radiotherapy, usually used for the treatment of tumours, was confirmed to be feasible, safe and effective in destroying abnormal tissue in heart by targeting high energy heavy ion beams at a specific area of the body precisely. In this study we will determine whether radiation ablation, can be used to destroy the thick heart muscle at the point of obstruction safely and effectively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years
* Drug-refractory symptomatic patients with HOCM
* Willing and able to give written informed consent

Exclusion Criteria:

* Enrolled in another clinical study.
* Patient unable to tolerate lying flat for one hour
* Pregnant Or Lactating Women
* With other contraindications for receive stereotactic ablative radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Safety of stereotactic ablative radiotherapy | 3 months
  The primary safety endpoint is defined as serious adverse events (SAEs) that are possibly/probably/definitely related to study treatment, based on previously published data for expected invasive alcohol septal-ablation procedures.

SECONDARY OUTCOMES:
Assessment of MACE endpoints | 1, 3, 6 and 12 months
  death, heart failure, myocardial infarction and stroke
Development of complete heart block, atrial or ventricular arrhythmias | 1, 3, 6 and 12 months
  diagnosis by electrocardiogram
Change in LVOT gradient | 1, 3, 6 and 12 months
  Assessed with transthoracic echocardiography
Change in exercise capacity | 1, 3, 6 and 12 months
  6 minute Walk Test
Change in LV wall thickness | 1, 3, 6 and 12 months
  Measured on echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Zhu Z, Liu J, Gao Y, Xiao Y, Fang Z, Liu Q, Liu X, Hu C, Ma F, Zeng M, Liu Z, Hu L, Liu N, Xiang F, Hu X, Huang L, Zhou S. Septal radioablation therapy for patients with hypertrophic obstructive cardiomyopathy: first-in-human study. Eur Heart J Open. 2023 May 23;3(3):oead052. doi: 10.1093/ehjopen/oead052. eCollection 2023 May. PMID 37503357